CLINICAL TRIAL: NCT01788423
Title: Evaluating Hearing Aid Service Delivery Models
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Larry Humes, Distinguished Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1111007504; R01DC011771 (NIH)
Record Dates: First submitted 2012-10-24; First posted 2013-02-11 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Presbycusis; Aging; Hearing Loss
Keywords: presbycusis; hearing aids
MeSH Terms: conditions — Presbycusis; Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Audiologist-Based (Experimental): Audiologist selects hearing aid for patient
  Interventions: Device: hearing aid
- Consumer Decides (Experimental): Consumer selects hearing aid
  Interventions: Device: hearing aid
- Placebo (Placebo Comparator): Patient fitted with hearing aid that is acoustically transparent.
  Interventions: Device: hearing aid

INTERVENTIONS:
Device: hearing aid — All subjects received hearing aids, some selected by audiologist, some selected by consumer, and some programmed as placebo devices.

SUMMARY:
The purpose of this study is to compare the outcomes for two different hearing-aid delivery models. In one model, the audiologist selects and fits the hearing aid and, in the other model, the consumer does this directly.

DETAILED DESCRIPTION:
The objectives of this study were to determine efficacy of hearing aids in older adults using audiology best practices, to evaluate the efficacy of an alternative over-the-counter (OTC) intervention, and to examine the influence of purchase price on outcomes for both service-delivery models. The design of this study was a single-site, prospective, double-blind placebo-controlled randomized trial with three parallel branches: (a) audiology best practices (AB), (b) consumer decides OTC model (CD), and (c) placebo devices (P). Outcome measures were obtained after a typical 6-week trial period with follow-up 4-week AB-based trial for those initially assigned to CD and P groups.

Older adults from the general community were recruited via newspaper and community flyers to participate at a university research clinic. Participants were adults, ages 55-79 years,with mild-to-moderate hearing loss. Intervention(s): All participants received the same highenddigital mini-behind-the-ear hearing aids fitted bilaterally.AB and P groups received best-practice services from audiologists; differing mainly in use of appropriate (AB) or placebo (P) hearing aid settings. CD participants self-selected their own pre-programmed hearing aids via an OTC model. Primary outcome measure was a 66-item self-report, Profile of Hearing Aid Performance/Benefit. Secondary outcome measure was the Connected Speech Test benefit.

ELIGIBILITY:
Inclusion Criteria: (for groups 1-4)

* 55-79 yrs of age
* Native English speaker
* no prior hearing aid use
* ability to read 18 point font

Exclusion Criteria: (for groups 1-3)

* hearing loss too severe or too mild for hearing aid
* middle-ear conductive pathology present
* asymmetrical hearing loss
* presence of dementia, Parkinson's disease, or other neurological disorder

Exclusion Criteria : (for groups 1-4)

- subject not interested in purchasing hearing aids

Ages: 55 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2012-11; Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry E. Humes, PhD, Principal Investigator — Indiana University
Locations (1):
- IU Department of Speech & Hearing Sciences, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, study forms, and final publication all available via Open Access publication in the American Journal of Audiology in March, 2017. De-identified individual data available from PI upon request.
Supporting Information: Study Protocol, ICF
Time Frame: Already available online with Open Access publication of the study in March, 2017.
Access Criteria: Open Access to protocol, study forms, and detailed results via publication in March, 2017. De-identified data available from investigator upon request.

REFERENCES:
- [Derived] Humes LE, Kinney DL, Main AK, Rogers SE. A Follow-Up Clinical Trial Evaluating the Consumer-Decides Service Delivery Model. Am J Audiol. 2019 Mar 15;28(1):69-84. doi: 10.1044/2018_AJA-18-0082. PMID 30938563
- [Derived] Humes LE, Rogers SE, Quigley TM, Main AK, Kinney DL, Herring C. The Effects of Service-Delivery Model and Purchase Price on Hearing-Aid Outcomes in Older Adults: A Randomized Double-Blind Placebo-Controlled Clinical Trial. Am J Audiol. 2017 Mar 1;26(1):53-79. doi: 10.1044/2017_AJA-16-0111. PMID 28252160

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial commenced November 2, 2012, and data collection ended August 31, 2016. Participants were recruited primarily by ads posted in the local newspapers and around the community. All testing of this volunteer sample took place in a university research clinic at Indiana University, Bloomington.
Pre-assignment Details: Of the 323 participants enrolled for assessment of eligibility, 135 were excluded because they did not meet inclusion criteria and 25 declined to participate, leaving 163 to be randomly allocated to one of the three intervention groups.
Period: Overall Study
Arm/Group | Audiologist-Based | Consumer Decides | Placebo
Started | 53 | 55 | 55
Completed | 53 | 51 (Four participants were unable to self-select hearing aids.) | 50 (Three people developed unrelated health problems and two were unable to fit/use hearing aids.)
Not Completed | 0 | 4 | 5
Not completed — See Comments in Completed (above) | 0 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Audiologist-Based | Consumer Decides | Placebo | Total
Number analyzed (Participants) | 53 | 51 | 50 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (5.6) | 68.0 (6.2) | 69.5 (6.7) | 69.1 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 16 | 67
  Male | 28 | 25 | 34 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 52 | 50 | 50 | 152
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 2 | 3
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 52 | 50 | 47 | 149
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants] — Midwestern United States based on residence reported.
  Participants
    United States | 53 | 51 | 50 | 154

OUTCOME MEASURES:

1. Primary Outcome: Profile of Hearing Aid Performance Benefit (PHAB)
Description: Change from unaided to aided performance on the Profile of Hearing Aid Performance with the difference in aided and unaided scores labeled Profile of Hearing Aid Benefit (PHAB), a self-report measure of benefit. The aided and unaided PHAP scores are proportions of time difficulties encountered in various listening situations. Low PHAP scores indicate less frequent difficulties. When subtracting aided from unaided PHAP scores, a positive PHAB score reflects less frequent problems when wearing a hearing aid compared to without. The range of possible PHAB scores are -1.0 to +1.0 with 0.0 indicating no difference between aided and unaided performance.
  There are seven subscales of the PHAP/PHAB and the scores reported are based on the arithmetic means of the five subscales that deal with speech communication, PHABglobal. These include the following subscale scores: EC (Ease of Communication), FT (Familiar Talkers), BN (Background Noise), Reverberation (RV) and Reduced Cues (RC).
Time Frame: two times: at hearing-aid fit and at 6-weeks post-fit
Measure: Mean (Standard Deviation); unit: Proportion of time had difficulties
Arm/Group | Audiologist-Based | Consumer Decides | Placebo
Number analyzed (Participants) | 53 | 51 | 50
Proportion of time had difficulties | 0.17 (0.12) | 0.12 (0.12) | 0.04 (0.10)

2. Secondary Outcome: Connected Speech Test (CST) Benefit
Description: A standardized speech-perception test, based on meaningful sentences and keyword scoring, the Connected Speech Test (CST) was administered unaided and aided. Each CST score represents the percentage of keywords (out of 50) repeated correctly following presentation via loudspeakers. Scores can range from 0 to 100% correct with higher scores indicating better speech perception. For the CST benefit scores reported below, unaided CST scores are subtracted from aided scores such that positive values represent better performance for aided than unaided listening. The possible range of CST benefit scores is -100 to +100 with 0 representing no difference between unaided and aided speech-perception performance.
Time Frame: two times: at hearing-aid fit and at 6-weeks post-fit
Measure: Mean (Standard Deviation); unit: Percentage of keywords correct
Arm/Group | Audiologist-Based | Consumer Decides | Placebo
Number analyzed (Participants) | 53 | 51 | 50
Percentage of keywords correct | 21.3 (19.4) | 26.6 (16.1) | 8.7 (21.2)

ADVERSE EVENTS:
Time Frame: 46 months
Arm/Group | Audiologist-Based | Consumer Decides | Placebo
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/51 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/51 | 0/50
Other Adverse Events (participants affected / at risk) | 0/53 | 0/51 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2012-11-02): https://cdn.clinicaltrials.gov/large-docs/23/NCT01788423/Prot_000.pdf